CLINICAL TRIAL: NCT06292572
Title: Clinical Characteristics and Surgical Outcomes of the Fellow Eye in Bilateral Retinal Detachments
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Professeur Jean-Baptiste CONART, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2024PI029
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Retinal Detachment
Keywords: retinal detachment; bilateral; vitrectomy
MeSH Terms: conditions — Retinal Detachment | interventions — Scleral Buckling; Predictive Value of Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initial Retinal Detachment: First of both eyes of the same patient that underwent retinal detachment repair
  Interventions: Procedure: Retinal Detachment Surgery
- Subsequent Retinal Detachment: Subsequent eye undergoing retinal detachment repair
  Interventions: Procedure: Retinal Detachment Surgery

INTERVENTIONS:
Procedure: Retinal Detachment Surgery — Retinal Detachment Surgery that consists in either Pars Plana Vitrectomy or Scleral Buckling or a combination of both techniques, and with or without use of intraocular tamponade
  Other Names: Pars plana Vitrectomy (PPV); Scleral Buckle (SB); PPV + SB

SUMMARY:
To assess the clinical features and the surgical outcomes of RD repair surgery of the fellow eye in bilateral retinal detachments

DETAILED DESCRIPTION:
Bilateral retinal detachment is a rare but sight-threatening disease, that can cause blindness and poor quality of life.

It has been proved that patients who suffer from RD in one eye have a considerably increased risk to subsequently develop an RD in the fellow eye.

It can be expected that patients who experienced a RD in one eye, tend to present sooner when experiencing a RD in the fellow eye, and thus have a greater visual and/or anatomical prognosis.

In this study, we aim to describe characteristics of bilateral RD and compare the initial and subsequent eye in terms of clinical preoperative features, surgical management, and anatomical and visual results.

ELIGIBILITY:
Inclusion Criteria:

* All patients that underwent retinal detachment repair surgery for bilateral sequential retinal detachment between January 2016 and December 2023 at the Nancy Regional and University Hospital Center (via pars plana vitrectomy or scleral buckling) and with a minimum of 6 month of post-operative follow-up after the last surgery.

Exclusion Criteria:

* Patients that underwent surgery at another facility
* Patients with a history of previous vitrectomy or
* Patients with a history of trauma from a penetrating injury or ruptured globe, retinal neovascular condition, hereditary vitreo-retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that underwent retinal detachment repair surgery for bilateral sequentiel retinal detachment between January 2016 and December 2023 at the Nancy Regional and University Hospital Center
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Rate of surgical success | 6 month after surgery
  Rate of succesful surgical repair of RD within the follow-up period

SECONDARY OUTCOMES:
Visual Acuity | 6 month after surgery
  LogMAR Visual acuity measured at the follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Conart, MD, PhD, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, Meurthe-et-Moselle, France

REFERENCES:
- [Background] Xu D, Belin PJ, Staropoli PC, Yannuzzi NA, Vangipuram G, Chiang A, Shah GK, Townsend JH, Ryan EH, Klufas MA. Clinical Outcomes in Sequential, Bilateral Rhegmatogenous Retinal Detachment: A Multicenter, Paired-Eye Analysis. Ophthalmol Retina. 2021 Aug;5(8):797-804. doi: 10.1016/j.oret.2020.11.002. Epub 2020 Nov 14. PMID 33197679
- [Background] Walia HS, Shah GK, Blinder KJ. Characteristics and outcomes of sequential rhegmatogenous retinal detachments. Ophthalmic Surg Lasers Imaging Retina. 2015 Apr;46(4):445-9. doi: 10.3928/23258160-20150422-07. PMID 25970865
- [Background] Mitry D, Singh J, Yorston D, Siddiqui MA, Murphy AL, Wright AF, Fleck BW, Campbell H, Charteris DG. The fellow eye in retinal detachment: findings from the Scottish Retinal Detachment Study. Br J Ophthalmol. 2012 Jan;96(1):110-3. doi: 10.1136/bjo.2010.194852. Epub 2011 Mar 3. PMID 21378003
- [Background] Radeck V, Schindler F, Helbig H, Gamulescu MA, Cvetkov Y, Barth T, Maerker D. Characteristics of Bilateral Retinal Detachment. Ophthalmologica. 2023;246(2):99-106. doi: 10.1159/000527625. Epub 2022 Oct 25. PMID 36282053
- [Background] Mastropasqua L, Carpineto P, Ciancaglini M, Falconio G, Gallenga PE. Treatment of retinal tears and lattice degenerations in fellow eyes in high risk patients suffering retinal detachment: a prospective study. Br J Ophthalmol. 1999 Sep;83(9):1046-9. doi: 10.1136/bjo.83.9.1046. PMID 10460773